CLINICAL TRIAL: NCT01848119
Title: Does a Perioperative Course of Gabapentin Improve Analgesia After Cesarean Delivery? A Randomised, Double-blind, Placebo Controlled Trial
Brief Title: Does a Perioperative Course of Gabapentin Improve Analgesia After Cesarean Delivery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-01
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Pain
Keywords: Gabapentin; Cesarean section
MeSH Terms: conditions — Pain | interventions — Gabapentin; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Active Comparator): Gabapentin 600mg, 1 dose preoperatively, followed by Gabapentin 200mg tid for 5 doses.
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): lactose capsules
  Interventions: Drug: lactose

INTERVENTIONS:
Drug: Gabapentin
  Other Names: Novo-gabapentin; Neurontin
  Arms: Gabapentin
Drug: lactose
  Arms: Placebo

SUMMARY:
Gabapentin has been very effective at treating pain after knee and hip operations, hysterectomies, and many other types of operations. A previous study at the investigators' hospital found that a single pre-operative dose of 600mg gabapentin produced a significant reduction in pain after cesarean section. However, 19% of patients complained of sedation. A subsequent study at the same institution looked to see if lowering the dose to 300mg would decrease pain scores whilst reducing the sedative side-effect seen in the first trial. The results were inconclusive but it provided valuable information to guide the design of this study.

The purpose of this study is to see whether a preoperative dose of gabapentin, followed by a 48 hour low-dose course will produce improvement in pain scores. This study will compare the efficacy of a peri-operative course of gabapentin (600mg one hour before the operation and 200mg every 8 hours for 2 days post-operatively) and a similar course of placebo in women undergoing Cesarean section. The investigators' hypothesis is that a course of gabapentin will result in decreased pain scores and increased satisfaction.

DETAILED DESCRIPTION:
Postoperative pain can have a significant negative impact on the physical and psychological health of both mother and child after cesarean delivery. Furthermore, severe postoperative pain may lead to persistent pain for many months. Therefore, optimal prevention and treatment of post cesarean pain is of paramount importance in women's health.

The current analgesic regimen most commonly used to manage pain after cesarean delivery includes neuraxial opioids, systemic acetaminophen and nonsteroidal anti-inflammatories, and systemic opioids for breakthrough pain. Although much improvement has been made with this regimen, pain scores assessment at 24 and 48 hours post cesarean delivery still show moderate pain, so further strategies to improve pain management are warranted.

Gabapentin has been shown to reduce pain scores and opioid consumption in the post-operative period in a variety of surgical settings such as hysterectomy and mastectomy. Studies have also shown a benefit in continuing the drug as a peri-operative course.

The use of gabapentin in cesarean deliveries is limited to 2 studies. The first trial at Mount Sinai Hospital found that a single dose of 600mg of gabapentin, administered preoperatively, significantly reduced the pain and increased the level of satisfaction of mothers who had delivered by cesarean section. There was however an increase in levels of sedation seen in those who received gabapentin and so a subsequent study was designed to see whether a reduced dose of 300mg could replicate the benefits shown without making mothers as drowsy. Unfortunately this study did not allow definitive conclusions to be drawn from the results as regards analgesic benefit, however the investigators did not observe an increase in sedation in patients receiving either 300 mg or 600 mg of gabapentin. Further studies are warranted to better define the role of gabapentin in this patient population.

The purpose of this study is to evaluate the efficacy of a preoperative dose of gabapentin followed by a short course of gabapentin in the first 48 hours post cesarean delivery, in the context of a multimodal analgesic regimen inclusive of intrathecal morphine and systemic NSAIDs, acetaminophen and opioids.

We hypothesize that this regimen will decrease VAS pains scores and increase maternal satisfaction post cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* All women aged 16 years and over with term singleton pregnancies undergoing elective cesarean delivery at Mount Sinai Hospital under spinal anesthesia, who have given pre-operative informed written consent will be eligible to participate in this study

Exclusion Criteria:

* Patients who have refused, are unable to give or have withdrawn consent
* Patients unable to communicate fluently in English
* Patients with American Society of Anesthesiologists (ASA) classification of 3 or greater
* Patients with history of epilepsy or chronic pain, or of use of anti-epileptic drugs or neuropathic analgesic drugs
* Patients with a history of opioid or intravenous drug abuse
* Patients with a known allergy or contra-indication to gabapentin, or to any other drugs used in this trial
* Patients who have refused spinal anaesthesia, or those in whom it is contra-indicated
* Patients with known congenital fetal abnormalities
* Patients who have taken antacid medication in the previous 24 hours

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 204 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
VAS score (VAS 0-100 mm) for maternal pain on movement at 24 hours after surgical incision. | 24 hours

SECONDARY OUTCOMES:
VAS score on movement at 48 hours after surgical incision | 48 hours
VAS scores at rest at 24 and 48 hours after surgical incision | 48 hours
Maternal satisfaction scores at 24 and 48 hours after surgical incision. | 48 hours
Opioid use in the first 48 hours after surgical incision | 48 hours
Time to first analgesic | 48 hours
  Time at which the patient requests any additional analgesic within the 48 hours after surgical incision.
Side effects; sedation, nausea, vomiting, dizziness, pruritis and difficulties balancing | 48 hours
  Patients exhibiting any sedation, nausea, vomiting, dizziness, pruritis and difficulties balancing in the 48 hours after surgical incision.
Neonatal apgar scores | 5 minutes
  Neonatal apgars scores at 1 and 5 minutes post delivery
Breastfeeding issues | 48 hours
  The presence of any difficulties breastfeeding that requires a lactation consult while in hospital.
NICU admission | 48 hours
  Any admissions to NICU of infants born to mothers participating in the study.
Anxiety level | 5 minutes
  Anxiety level recorded on a Numeric Rating Scale of 0-10 (0 = "no anxiety", 10 = "the most severe anxiety possible"), prior to surgery.
Pain Catastrophizing Scale (PCS) questionnaire. | 15 minutes
  The PCS questionnaire is a pain research tool that examines a subject's pain related psychology.

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada